CLINICAL TRIAL: NCT05871229
Title: Prevention of Dental Implant Diseases: Early Diagnosis and Monitoring in Clinical Work and Enhanced Oral Health Maintenance at Home
Brief Title: Prevention of Dental Implant Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanna Lähteenmäki (Industry)
Collaborators: University of Helsinki (Other); Koite Health Oy (Industry); Hammasklinikka Kruunu (Unknown)
Responsible Party: Sponsor-Investigator, Hanna Lähteenmäki, PhD, Dental Hygienist, Koite Health Oy
Organization: Koite Health Oy (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IS-TRE
Record Dates: First submitted 2023-05-03; First posted 2023-05-23 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Peri-Implantitis
Keywords: Peri-implant disease; aMMP-8; Antibacterial photodynamic therapy (aBPT); Oral hygiene
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Investigator
Masking Description: Participants will be randomized at the end of baseline visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Lumoral and standard treatment
  Interventions: Device: Lumoral Treatment; Other: Standard treatment for peri-implantitis
- Control group (Other): Standard treatment only
  Interventions: Other: Standard treatment for peri-implantitis

INTERVENTIONS:
Device: Lumoral Treatment — Photodynamic antibacterial dual-light device with a marker substance
  Arms: Study group
Other: Standard treatment for peri-implantitis — Standard treatment for peri-implantitis as per international, national and clinic guidelines

SUMMARY:
The aim of this study is to determine the effect of regular antibacterial photodynamic Lumoral® treatment on gingival health and plaque volume, and anti-inflammatory effect of daily double light therapy on implant teeth. The study will use a medical device containing a light-activated Lumorinse® mouthwash and a Lumoral® light activator.

DETAILED DESCRIPTION:
The hypothesis is that antibacterial photodynamic therapy improves tissue health by reducing inflammation without any side effect.

Study participants will be invited from a dental clinic in Tampere, Finland, from the patients of an oral hygienist's office. Participants will be randomized to the treatment and control groups using the closed envelope method. Participants in the treatment group will receive Lumoral® treatment according to the manufacturer's protocol, once daily for 10 min for 15 days and then twice daily for 15 days.

ELIGIBILITY:
Inclusion Criteria:

* One or more dental implants
* Diagnosis of peri-implantitis
* Challenges in keeping high self-care oral care standards
* Over 25 years of age

Exclusion Criteria:

- Any antibiotic medication within 6 months prior to study participation

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Active matrix metalloproteinase 8 (aMMP-8) | 30 days
  Change in periodontal inflammation marker aMMP-8

SECONDARY OUTCOMES:
Bleeding on probing (BOP) | 30 days
  Improvement in bleeding on probing (BOP)
  A full-mouth assessment at six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual, lingual, distolingual) Gingival bleeding is considered as positive if bleeding occurs within 15 seconds after gentle probing with a probe at the sulcus Dichotomous scoring to each site of the tooth as bleeding "1 present" and "0 absent" BOP is reported as the percentage (%) of sites with positive findings Calculation formula: number of bleeding sites/ 6 times number of teeth
Visible plaque index (VPI) | 30 days
  Change in visible plaque index

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Lähteenmäki, Doctor, Principal Investigator — Hammasklinikka Kruunu
Locations (1):
- Hammasklinikka Kruunu Oy, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhir S, Mahesh L, Kurtzman GM, Vandana KL. Peri-implant and periodontal tissues: a review of differences and similarities. Compend Contin Educ Dent. 2013 Jul-Aug;34(7):e69-75. PMID 24428439
- [Background] Matsubara T, Kusuzaki K, Matsumine A, Satonaka H, Shintani K, Nakamura T, Uchida A. Methylene blue in place of acridine orange as a photosensitizer in photodynamic therapy of osteosarcoma. In Vivo. 2008 May-Jun;22(3):297-303. PMID 18610739
- [Background] Raisanen IT, Heikkinen AM, Nwhator SO, Umeizudike KA, Tervahartiala T, Sorsa T. On the diagnostic discrimination ability of mouthrinse and salivary aMMP-8 point-of-care testing regarding periodontal health and disease. Diagn Microbiol Infect Dis. 2019 Dec;95(4):114871. doi: 10.1016/j.diagmicrobio.2019.114871. Epub 2019 Jul 26. PMID 31473032
- [Background] Salvi GE, Zitzmann NU. The effects of anti-infective preventive measures on the occurrence of biologic implant complications and implant loss: a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:292-307. doi: 10.11607/jomi.2014suppl.g5.1. PMID 24660205
- [Background] Schwarz F, Becker K, Sager M. Efficacy of professionally administered plaque removal with or without adjunctive measures for the treatment of peri-implant mucositis. A systematic review and meta-analysis. J Clin Periodontol. 2015 Apr;42 Suppl 16:S202-13. doi: 10.1111/jcpe.12349. PMID 25496187
- [Background] Shinwari MS, Tanwir F, Hyder PR, Bin Saeed MH. Host modulation therapeutics in periodontics: role as an adjunctive periodontal therapy. J Coll Physicians Surg Pak. 2014 Sep;24(9):676-84. PMID 25233975
- [Background] Smeets R, Henningsen A, Jung O, Heiland M, Hammacher C, Stein JM. Definition, etiology, prevention and treatment of peri-implantitis--a review. Head Face Med. 2014 Sep 3;10:34. doi: 10.1186/1746-160X-10-34. PMID 25185675
- [Background] Sorsa T, Gieselmann D, Arweiler NB, Hernandez M. A quantitative point-of-care test for periodontal and dental peri-implant diseases. Nat Rev Dis Primers. 2017 Sep 14;3:17069. doi: 10.1038/nrdp.2017.69. No abstract available. PMID 28905941
- [Background] Sorsa T, Hernandez M, Leppilahti J, Munjal S, Netuschil L, Mantyla P. Detection of gingival crevicular fluid MMP-8 levels with different laboratory and chair-side methods. Oral Dis. 2010 Jan;16(1):39-45. doi: 10.1111/j.1601-0825.2009.01603.x. Epub 2009 Jul 8. PMID 19627514
- [Background] Sorsa T, Tjaderhane L, Salo T. Matrix metalloproteinases (MMPs) in oral diseases. Oral Dis. 2004 Nov;10(6):311-8. doi: 10.1111/j.1601-0825.2004.01038.x. PMID 15533204
- [Background] Suarez-Lopez Del Amo F, Yu SH, Wang HL. Non-Surgical Therapy for Peri-Implant Diseases: a Systematic Review. J Oral Maxillofac Res. 2016 Sep 9;7(3):e13. doi: 10.5037/jomr.2016.7313. eCollection 2016 Jul-Sep. PMID 27833738
- [Background] Terheyden H, Stadlinger B, Sanz M, Garbe AI, Meyle J. Inflammatory reaction - communication of cells. Clin Oral Implants Res. 2014 Apr;25(4):399-407. doi: 10.1111/clr.12176. Epub 2013 Apr 21. PMID 23600659
- See also: Hentilä, J. et al. (2021). Dual-Light Photodynamic Therapy Effectively Eliminates Streptococcus Oralis Biofilms. Journal of Pharmacy & Pharmaceutical Sciences, 24 — https://journals.library.ualberta.ca/jpps/index.php/JPPS/article/view/32084
- See also: Kilian, M. et al. (2016). The oral microbiome - An update for oral healthcare professionals. British Dental Journal, 221(10). — https://www.nature.com/articles/sj.bdj.2016.865
- See also: Kormi, I et al. (2014) The effect of prolonged systemic doxycycline therapy on serum tissue degrading proteinases in coronary bypass patients: a randomized, double-masked, placebo-controlled clinical trial. Inflammation Research, 63(5), 329-334 — https://link.springer.com/article/10.1007/s00011-013-0704-2
- See also: Nikinmaa, S., et al. (2020). Dual-light photodynamic therapy administered daily provides a sustained antibacterial effect on biofilm and prevents Streptococcus mutans adaptation. PloS One, 15(5). — https://doi.org/10.1371/journal.pone.0232775